CLINICAL TRIAL: NCT01428531
Title: Special Drug Use Investigation for Arixtra® (Fondaparinux) Venous Thromboembolism Treatment
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115489
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Ataxia
MeSH Terms: conditions — Ataxia | interventions — Fondaparinux

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients prescribed fondaparinux
  Interventions: Drug: Fondaparinux Sodium

INTERVENTIONS:
Drug: Fondaparinux Sodium

SUMMARY:
The purpose of this post-marketing surveillance study is to collect and assess information on safety and efficacy of fondaparinux injection in patients with venous thromboembolism (VTE).

("Arixtra" is a trademark of the GlaxoSmithKline group of companies.)

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute pulmonary thromboembolism or acute deep venous thrombosis
* Fondaparinux injection must be prescribed for the first time

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese patients with acute pulmonary thromboembolism or acute deep venous thrombosis
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse drug reaction | 3 months
Number of patients with any serious adverse event | 3 months
Number of patients with any hemorrhagic adverse event | 3 months
Presence or absence of reoccurrence of VTE | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline